CLINICAL TRIAL: NCT07138118
Title: Effects of an Individualized Blood Flow Restriction Training Combined With a Cognitive-Motor Dual Task Intervention on Lower Limb Strength, Gait Ability, and Fall Stability in Subacute Stroke Patients: A Randomized Controlled Trial
Brief Title: Study of Blood Flow Restriction and Cognitive-Motor Dual Task Training to Improve Strength, Gait, and Balance in People With Subacute Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sahmyook University (Other)
Responsible Party: Principal Investigator, Seonghwan Kim, Principal Investigator, MSc Candidate, Department of Physical Therapy, Sahmyook University, Sahmyook University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SYU 2025-06-027-001
Record Dates: First submitted 2025-08-15; First posted 2025-08-22 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-09

CONDITIONS: Subacute Stroke
Keywords: Subacute Stroke; BFR; Dual Task Training; Gait; Balance; Muscle Strength; Falls Efficacy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: BFR + Dual Task (Experimental): Participants in this group will perform cognitive-motor dual task training while wearing blood flow restriction (BFR) cuffs set at 40% of their individualized arterial occlusion pressure (AOP). The training consists of three sessions per week for five weeks. Each session lasts 40 minutes and includes tasks such as forward walking, obstacle crossing, and seated-to-stand with concurrent verbal fluency or serial subtraction tasks.
  Interventions: Behavioral: Blood Flow Restriction + Dual Task Training
- Active Comparator: Dual Task Only (Active Comparator): Participants in this group will perform the same cognitive-motor dual task training as the experimental group but without blood flow restriction. The training will also be conducted three times per week for five weeks, with each session lasting 40 minutes. Tasks include walking and obstacle navigation combined with verbal fluency or serial subtraction exercises.
  Interventions: Behavioral: Dual Task Training Only

INTERVENTIONS:
Behavioral: Blood Flow Restriction + Dual Task Training — Participants will undergo lower limb resistance and gait training while wearing blood flow restriction cuffs at 40% of their individualized arterial occlusion pressure. Tasks include walking, sit-to-stand, and obstacle crossing combined with verbal fluency or serial subtraction. Training is performed 3 times per week for 5 weeks.
  Other Names: BFR-DT; Individualized BFR
  Arms: Experimental: BFR + Dual Task
Behavioral: Dual Task Training Only — Participants will perform the same cognitive-motor dual task training without blood flow restriction. Tasks include forward walking, obstacle crossing, and sit-to-stand exercises with concurrent cognitive tasks such as verbal fluency or serial subtraction. Training is performed 3 times per week for 5 weeks.
  Other Names: Dual Task Gait Training; DT
  Arms: Active Comparator: Dual Task Only

SUMMARY:
This study aims to evaluate the effects of individualized blood flow restriction (BFR) training combined with cognitive-motor dual task intervention on lower limb muscle strength, gait ability, and fall stability in patients with subacute stroke. A total of 28 participants will be randomly assigned to either the experimental group (BFR + dual task training) or the control group (dual task only). The intervention will last for 5 weeks, with training sessions conducted three times per week, each lasting 40 minutes. The primary outcome is lower limb strength measured by the Five Times Sit-to-Stand Test. Secondary outcomes include gait ability (10-Meter Walk Test and Functional Gait Assessment) and fall stability (Timed Up and Go Test and Korean version of the Falls Efficacy Scale-International). This study seeks to verify whether combining low-pressure BFR training (40% of arterial occlusion pressure) with dual task training can be a clinically effective strategy for improving motor and cognitive function in individuals with subacute stroke.

DETAILED DESCRIPTION:
Subacute stroke is defined as the period between 7 days and 6 months after stroke onset, a critical window during which neuroplasticity and functional recovery are highly active. During this phase, individualized and task-specific interventions can enhance motor recovery. Blood flow restriction (BFR) training is a promising low-load exercise modality that induces physiological effects similar to high-intensity training by restricting venous return using a proximal cuff. Studies suggest that BFR training at 40% of arterial occlusion pressure (AOP) can safely stimulate muscle hypertrophy and strength, particularly in populations with limited exercise capacity, such as stroke survivors.

Additionally, dual task training, which combines motor and cognitive tasks, has been shown to improve executive function and gait performance by increasing prefrontal cortex activity. While each approach has independent benefits, the combination of peripheral muscle activation through BFR and central stimulation via cognitive-motor dual tasks may provide synergistic effects on functional recovery.

This randomized controlled trial will compare an intervention group receiving BFR training (40% AOP) with concurrent dual task gait training to a control group performing the same cognitive-motor dual tasks without BFR. Both groups will train three times per week for 5 weeks. Outcome measures will assess changes in lower limb strength, gait ability, and fall stability before and after the intervention. The study also addresses safety and standardization concerns in BFR application by using pulse oximeter-based AOP measurement protocols.

By providing evidence on the efficacy and safety of combining BFR and dual-task training in subacute stroke rehabilitation, this study aims to contribute to the development of individualized, clinically applicable intervention strategies.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with subacute stroke within 1 to 6 months after onset
* Able to walk at least 10 meters, with or without assistive devices
* Modified Ashworth Scale score less than 1
* Korean Mini-Mental State Examination (K-MMSE) score of 24 or higher

Exclusion Criteria:

* History of psychiatric disorders or cognitive impairment
* Presence of peripheral neuropathy
* Resting systolic blood pressure ≥160 mmHg or diastolic blood pressure ≥100 mmHg despite medication
* Diagnosis of heart failure or unstable angina
* History of bypass surgery within the past 3 months
* Serious musculoskeletal disorders affecting gait (e.g., amputation, fracture)

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2025-09-08 (Actual); Primary Completion 2025-10-17 (Actual); Study Completion 2025-11-11 (Actual)

PRIMARY OUTCOMES:
5 Times Sit-to-Stand Test (5STS) | Baseline and after 5 weeks of intervention
  Lower limb strength will be assessed using the Five Times Sit-to-Stand Test. A shorter time indicates better performance.

SECONDARY OUTCOMES:
10-Meter Walk Test (10MWT) | Baseline and after 5 weeks of intervention
  Walking speed (m/s) will be measured over a middle 10-meter segment of a 14-meter walking path. Higher values indicate better performance.
Timed Up and Go Test (TUG) | Baseline and after 5 weeks of intervention
  Shorter completion time on the TUG indicates improved functional balance and mobility.
Korean Version of Falls Efficacy Scale - International (KFES-I) | Baseline and after 5 weeks of intervention
  KFES-I assesses confidence in avoiding falls during daily activities. Lower scores indicate higher confidence.
Functional Gait Assessment (FGA) | Baseline and after 5 weeks of intervention
  The FGA is a 10-item test that assesses postural stability during various walking tasks. Higher scores indicate better functional gait and balance.

CONTACTS AND LOCATIONS:
Overall Officials: Seungwon Lee, PhD, Principal Investigator — Sahmyook University
Locations (1):
- Sahmyook University, Seoul, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Liu YC, Yang YR, Tsai YA, Wang RY. Cognitive and motor dual task gait training improve dual task gait performance after stroke - A randomized controlled pilot trial. Sci Rep. 2017 Jun 22;7(1):4070. doi: 10.1038/s41598-017-04165-y. PMID 28642466
- [Result] Ahmed I, Mustafaoglu R, Erhan B. The effects of low-intensity resistance training with blood flow restriction versus traditional resistance exercise on lower extremity muscle strength and motor functionin ischemic stroke survivors: a randomized controlled trial. Top Stroke Rehabil. 2024 May;31(4):418-429. doi: 10.1080/10749357.2023.2259170. Epub 2023 Sep 19. PMID 37724785